CLINICAL TRIAL: NCT03638609
Title: The Effect of Intra Aortic Balloon Pump Early Insertion on Mortality in Post Cardiac Arrest Patients With Acute Coronary Syndrome
Brief Title: The Effect of IABP Early Insertion on Mortality in Post Cardiac Arrest Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Isman Firdaus, MD, Interventional Cardiologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IABP17
Record Dates: First submitted 2018-08-09; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Post-Cardiac Arrest Syndrome
Keywords: IABP; Post-Cardiac Arrest Syndrome; Beclin-1; Caspase-3; Mortality
MeSH Terms: conditions — Post-Cardiac Arrest Syndrome; Spinocerebellar Ataxias | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Group of patients not receiving IABP
- Intra Aortic Balloon Pump (Experimental): Group of patients receiving Intra Aortic Balloon Pump in 3 hours after ROSC (early insertion of IABP)
  Interventions: Device: Intra Aortic Balloon Pump

INTERVENTIONS:
Device: Intra Aortic Balloon Pump — Intra Aortic Balloon Pump (IABP) is a circulatory mechanical support device, placed in descending aorta, distally from left subclavian artery and proximally from renal artery. IABP works with counterpulsation concept, synchronized with heart cycle. It is indicated as supportive therapy for patients undergoing revascularization, cardiogenic shock and mechanical complication.
  Balloon dilatation during dyastolic phase increasing dyastolic pressure in aorta, improving coronary vascularization and myocardial oxygen supply. In systolic phase, the balloon deflates, reducing the left ventricle afterload hence decreasing myocardial oxygen demand.
  Other Names: IABP
  Arms: Intra Aortic Balloon Pump

SUMMARY:
The prevalence of cardiac arrests is still high worldwide. Despite the return of spontaneous circulation (ROSC), mortality and morbidity in post cardiac arrest patients is reported high. Comprehensive management is essential in treating patients with post cardiac arrest syndrome. Adequate circulatory stability is achieved with fluid therapy, vasoactive drug therapy, and consideration of mechanical support. Intra-Aortic Ballon Pump (IABP) is one of the most feasible and available mechanical support in developing countries including Indonesia.

There are several benefits of IABP reported in acute myocardial infarction complicated with cardiogenic shock. Nevertheless, the IABP-SHOCK II study revealed contradictive result which is IABP support was not improving mortality in acute myocardial infarction complicated with cardiogenic shock after revascularization. Other study, Korean Acute Myocardial Infarction Registry (KAMIR), also reported no benefits of IABP support in cardiogenic shock patients. But, the study the investigators mentioned earlier is a registry study, attributed to selection bias and several confounding factors resulting mismatch in population. There are no consideration to IABP time of initiation and duration of use in both studies.

The Investigator is aiming to prove the early insertion of IABP to a better outcome compared with the absence of early IABP. The objective of the study is to assess mortality in post cardiac arrest syndrome patients with early insertion of IABP support. A total of 102 subjects will be enrolled in this study, divided into IABP and non-IABP group. The primary outcome is in-hopital-mortality, and various indicators in the pathomechanisme of post cardiac arrest syndrome will be measured in 30 minutes and 6 hours after ROSC. Effective lactate clearance, IL-6, Beclin-1, Caspase-3, a-vO2 diff, and ScvO2, cardiac output, VTI, TAPSE and ejection fraction will be measured and analized between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 and less than 75 years.
2. Post cardiac arrest syndrome patients with decreased level of consciousness (cerebral performance categories (CPC) more than 1) and hypotension (systolic blood pressure less than 100)
3. Experiencing successful cardiac rescucitation following cardiac arrest

Exclusion Criteria:

1. History of stroke (based on interview)
2. Unequal pupil
3. Previous use of IABP
4. Aorta regurgitation
5. Brugada syndrome and congenital long QT

Drop-out Criteria:

1. Participants who died before IABP insertion
2. The family requests for a termination of treatment.
3. Anemia caused by bleeding with hemoglobin decrement by >3 gr/dL
4. Ankle brachial index(ABI) less than 0,8

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-10-23 (Estimated); Study Completion 2018-11-23 (Estimated)

PRIMARY OUTCOMES:
In-Hospital Mortality | 30 days
  Mortality of patients during the hospitalization receiving early insertion IABP

CONTACTS AND LOCATIONS:
Overall Officials: Isman Firdaus, MD, Principal Investigator — National Cardiovascular Center Harapan Kita Hospital Indonesia
Locations (1):
- National Cradiovascular Center Harapan Kita Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams JA, Uryash A, Nadkarni V, Berg RA, Lopez JR. Whole body periodic acceleration (pGz) preserves heart rate variability after cardiac arrest. Resuscitation. 2016 Feb;99:20-5. doi: 10.1016/j.resuscitation.2015.11.018. Epub 2015 Dec 12. PMID 26690649
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Stub D, Bernard S, Duffy SJ, Kaye DM. Post cardiac arrest syndrome: a review of therapeutic strategies. Circulation. 2011 Apr 5;123(13):1428-35. doi: 10.1161/CIRCULATIONAHA.110.988725. No abstract available. PMID 21464058
- [Background] Firdaus I. Registry of Acute and Intensive Cardiovascular Care on Outcome (RAICOM) in National Cardiovascular Center Harapan Kita Indonesia. 2016.
- [Background] iSTEMI (Indonesia STEMI). 2016
- [Background] Jentzer JC, Chonde MD, Dezfulian C. Myocardial Dysfunction and Shock after Cardiac Arrest. Biomed Res Int. 2015;2015:314796. doi: 10.1155/2015/314796. Epub 2015 Sep 2. PMID 26421284
- [Background] Mongardon N, Dumas F, Ricome S, Grimaldi D, Hissem T, Pene F, Cariou A. Postcardiac arrest syndrome: from immediate resuscitation to long-term outcome. Ann Intensive Care. 2011 Nov 3;1(1):45. doi: 10.1186/2110-5820-1-45. PMID 22053891
- [Background] Pellis T, Sanfilippo F, Ristagno G. The optimal hemodynamics management of post-cardiac arrest shock. Best Pract Res Clin Anaesthesiol. 2015 Dec;29(4):485-95. doi: 10.1016/j.bpa.2015.10.002. Epub 2015 Oct 14. PMID 26670819
- [Background] He C, Levine B. The Beclin 1 interactome. Curr Opin Cell Biol. 2010 Apr;22(2):140-9. doi: 10.1016/j.ceb.2010.01.001. Epub 2010 Jan 22. PMID 20097051
- [Background] Kang R, Zeh HJ, Lotze MT, Tang D. The Beclin 1 network regulates autophagy and apoptosis. Cell Death Differ. 2011 Apr;18(4):571-80. doi: 10.1038/cdd.2010.191. Epub 2011 Feb 11. PMID 21311563
- [Background] Green DR, Llambi F. Cell Death Signaling. Cold Spring Harb Perspect Biol. 2015 Dec 1;7(12):a006080. doi: 10.1101/cshperspect.a006080. PMID 26626938
- [Background] McIlwain DR, Berger T, Mak TW. Caspase functions in cell death and disease. Cold Spring Harb Perspect Biol. 2013 Apr 1;5(4):a008656. doi: 10.1101/cshperspect.a008656. PMID 23545416
- [Background] Brentnall M, Rodriguez-Menocal L, De Guevara RL, Cepero E, Boise LH. Caspase-9, caspase-3 and caspase-7 have distinct roles during intrinsic apoptosis. BMC Cell Biol. 2013 Jul 9;14:32. doi: 10.1186/1471-2121-14-32. PMID 23834359
- [Background] Porter AG, Janicke RU. Emerging roles of caspase-3 in apoptosis. Cell Death Differ. 1999 Feb;6(2):99-104. doi: 10.1038/sj.cdd.4400476. PMID 10200555
- [Background] Jahania SM, Sengstock D, Vaitkevicius P, Andres A, Ito BR, Gottlieb RA, Mentzer RM Jr. Activation of the homeostatic intracellular repair response during cardiac surgery. J Am Coll Surg. 2013 Apr;216(4):719-26; discussion 726-9. doi: 10.1016/j.jamcollsurg.2012.12.034. Epub 2013 Feb 13. PMID 23415552
- [Background] Kassiotis C, Ballal K, Wellnitz K, Vela D, Gong M, Salazar R, Frazier OH, Taegtmeyer H. Markers of autophagy are downregulated in failing human heart after mechanical unloading. Circulation. 2009 Sep 15;120(11 Suppl):S191-7. doi: 10.1161/CIRCULATIONAHA.108.842252. PMID 19752367
- [Background] de Jonge N, van Wichen DF, van Kuik J, Kirkels H, Lahpor JR, Gmelig-Meyling FH, van den Tweel JG, de Weger RA. Cardiomyocyte death in patients with end-stage heart failure before and after support with a left ventricular assist device: low incidence of apoptosis despite ubiquitous mediators. J Heart Lung Transplant. 2003 Sep;22(9):1028-36. doi: 10.1016/s1053-2498(02)01160-9. PMID 12957613
- [Background] Prescimone T, Masotti S, D'Amico A, Caruso R, Cabiati M, Caselli C, Viglione F, Verde A, Del Ry S, Giannessi D. Cardiac molecular markers of programmed cell death are activated in end-stage heart failure patients supported by left ventricular assist device. Cardiovasc Pathol. 2014 Sep-Oct;23(5):272-82. doi: 10.1016/j.carpath.2014.04.003. Epub 2014 Apr 13. PMID 24856512
- [Background] Lazzeri C, Valente S, Chiostri M, Gensini GF. Clinical significance of lactate in acute cardiac patients. World J Cardiol. 2015 Aug 26;7(8):483-9. doi: 10.4330/wjc.v7.i8.483. PMID 26322188
- [Background] Andersen LW, Mackenhauer J, Roberts JC, Berg KM, Cocchi MN, Donnino MW. Etiology and therapeutic approach to elevated lactate levels. Mayo Clin Proc. 2013 Oct;88(10):1127-40. doi: 10.1016/j.mayocp.2013.06.012. PMID 24079682
- [Background] Englehart MS, Schreiber MA. Measurement of acid-base resuscitation endpoints: lactate, base deficit, bicarbonate or what? Curr Opin Crit Care. 2006 Dec;12(6):569-74. doi: 10.1097/MCC.0b013e328010ba4f. PMID 17077689
- [Background] Mullner M, Sterz F, Domanovits H, Behringer W, Binder M, Laggner AN. The association between blood lactate concentration on admission, duration of cardiac arrest, and functional neurological recovery in patients resuscitated from ventricular fibrillation. Intensive Care Med. 1997 Nov;23(11):1138-43. doi: 10.1007/s001340050470. PMID 9434919
- [Background] Donnino MW, Miller J, Goyal N, Loomba M, Sankey SS, Dolcourt B, Sherwin R, Otero R, Wira C. Effective lactate clearance is associated with improved outcome in post-cardiac arrest patients. Resuscitation. 2007 Nov;75(2):229-34. doi: 10.1016/j.resuscitation.2007.03.021. Epub 2007 Jun 20. PMID 17583412
- [Background] Lee TR, Kang MJ, Cha WC, Shin TG, Sim MS, Jo IJ, Song KJ, Jeong YK, Cho JH. Better lactate clearance associated with good neurologic outcome in survivors who treated with therapeutic hypothermia after out-of-hospital cardiac arrest. Crit Care. 2013 Oct 31;17(5):R260. doi: 10.1186/cc13090. PMID 24172276
- [Background] Cocchi MN, Miller J, Hunziker S, Carney E, Salciccioli J, Farris S, Joyce N, Zimetbaum P, Howell MD, Donnino MW. The association of lactate and vasopressor need for mortality prediction in survivors of cardiac arrest. Minerva Anestesiol. 2011 Nov;77(11):1063-71. Epub 2011 May 11. PMID 21597442
- [Background] Shinozaki K, Oda S, Sadahiro T, Nakamura M, Hirayama Y, Watanabe E, Tateishi Y, Nakanishi K, Kitamura N, Sato Y, Hirasawa H. Blood ammonia and lactate levels on hospital arrival as a predictive biomarker in patients with out-of-hospital cardiac arrest. Resuscitation. 2011 Apr;82(4):404-9. doi: 10.1016/j.resuscitation.2010.10.026. Epub 2011 Jan 11. PMID 21227564
- [Background] Kim HK, Jeong MH, Ahn Y, Sim DS, Chae SC, Kim YJ, Hur SH, Seong IW, Hong TJ, Choi DH, Cho MC, Kim CJ, Seung KB, Jang YS, Rha SW, Bae JH, Cho JG, Park SJ; other Korea Acute Myocardial Infarction Registry Investigators. Clinical outcomes of the intra-aortic balloon pump for resuscitated patients with acute myocardial infarction complicated by cardiac arrest. J Cardiol. 2016 Jan;67(1):57-63. doi: 10.1016/j.jjcc.2015.04.007. Epub 2015 May 14. PMID 25982668
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, de Waha A, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Lauer B, Bohm M, Ebelt H, Schneider S, Werdan K, Schuler G; Intraaortic Balloon Pump in cardiogenic shock II (IABP-SHOCK II) trial investigators. Intra-aortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock (IABP-SHOCK II): final 12 month results of a randomised, open-label trial. Lancet. 2013 Nov 16;382(9905):1638-45. doi: 10.1016/S0140-6736(13)61783-3. Epub 2013 Sep 3. PMID 24011548
- [Background] Dharma S, Dakota I, Firdaus I, Wardeh AJ, Jukema JW. The Use of Intra-aortic Balloon Pump in a Real-World Setting: A Comparison between Survivors and Nonsurvivors from Acute Coronary Syndrome Treated with IABP. The Jakarta Acute Coronary Syndrome Registry. Int J Angiol. 2013 Dec;22(4):213-22. doi: 10.1055/s-0033-1348884. PMID 24436615

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03638609/Prot_SAP_ICF_000.pdf